CLINICAL TRIAL: NCT05704101
Title: Influence of Nasal High-flow Therapy (NHFT) on Ventilation and Sympathetic Drive in Patients With Asthma
Brief Title: NHFT Effects on Symptatheic Drive of Asthma Patients
Acronym: MSNA in Asthma
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: CTCA 22-274
Record Dates: First submitted 2023-01-06; First posted 2023-01-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma patients (n=20) out of them 10 with mild, controlled and 10 with severe, uncontrolled asthma: * Assessments of the SNA-axis. For this, HRV and dBPV will be analyzed using a 3-lead ECG and a continuous non-invasive arterial blood pressure signal. HRV and dBPV will be computed and presented as the high frequency , low frequency , their relative ratio (LF/HF), and the very low frequency component for both.
  * MSNA will be recorded via a tungsten microelectrode placed in the peroneal nerve.
  * NHFT at a flow rate of 20/30/40 liters/minute for 30 minutes respectively, with breaks of 15 minutes for all physiological variables to return to baseline.
  * OSA severity: defined as apnoea-hypopnoea index [AHI] >15/h and obstructive apnoea index [OAI] >5/h
  * Determination of PH and right HF severity (TAPSE ≤14 mm) and pulmonary arterial pressure (PAsys) using TTE.
  * Comprehensive lung function and inspiratory muscle strength and function testing as described previously by our group.
  * Assessment of systemic inflammation in blood samples.
- Controls (n=10) (and in a group of healthy controls [2:1] matched for age, sex and BMI).: * Assessments of the SNA-axis. For this, HRV and dBPV will be analyzed using a 3-lead ECG and a continuous non-invasive arterial blood pressure signal. HRV and dBPV will be computed and presented as the high frequency , low frequency , their relative ratio (LF/HF), and the very low frequency component for both.
  * MSNA will be recorded via a tungsten microelectrode placed in the peroneal nerve.
  * NHFT at a flow rate of 20/30/40 liters/minute for 30 minutes respectively, with breaks of 15 minutes for all physiological variables to return to baseline.
  * OSA severity: defined as apnoea-hypopnoea index [AHI] >15/h and obstructive apnoea index [OAI] >5/h
  * Determination of PH and right HF severity (TAPSE ≤14 mm) and pulmonary arterial pressure (PAsys) using TTE.
  * Comprehensive lung function and inspiratory muscle strength and function testing as described previously by our group.
  * Assessment of systemic inflammation in blood samples.

SUMMARY:
The project will be pursued in our respiratory, autonomic nervous system physiology laboratory (Respiratory, autonomic nervous system physiology laboratory, Department of Pneumology and Intensive Care Medicine, RWTH Aachen University Hospital).

Overactivity of the sympathetic nerve activity (SNA) axis with "centrally" increased heart rate and peripheral vasoconstriction is a known phenomenon in patients with systolic heart failure (HF) and has recently been described in patients with primary lung diseases as in chronic obstructive pulmonary disease (COPD) and pulmonary hypertension (PH). Comprehensive studies investigating sympathetic drive in Asthma as one of the major pulmonary diseases are still lacking. Furthermore, the intention of this study is to determine the impact of Nasal High Flow Therapy (NHFT) on SNA and assess respiratory muscle function using state-of-the-art techniques.

DETAILED DESCRIPTION:
Asthma, being one of the major pulmonary diseases affects roughly 300 million people worldwide. This disease leads to airflow obstruction within the lung following chronic inflammation of the respiratory tract, which results in a wide range of symptoms. Overactivity of SNA has been already linked to patients with systolic heart failure and COPD. The investigators postulate that similar pathomechanism is prevalent in Asthma which leads to an overactivity of SNA.

Nasal High Flow Therapy (NHFT) is a recently developed form of oxygen therapy that delivers heated and humidified high-flow oxygen and gas mix through a nasal cannula. In comparison to conventional oxygen therapy, NHFT has been proven substantially beneficial due to additional effects like decreased oxygen dilution, increased FRC, dead space washout with CO2 removal, increased mucociliary function and generation of positive end-expiratory pressure (PEEP) which lead to significantly improved breathing mechanics often preventing the need for invasive machine ventilation (IMV) in various acute diseases. Furthermore, these mechanisms lead to the bronchodilation of small airways in primary obstructive pulmonary diseases like COPD. Positive benefits of NHFT, not only during an acute exacerbation but also with long-term stable disease have been already established in COPD. Similar effects could be expected in bronchial Asthma characterized by obstruction of small airways.

Thus, using a comprehensive, multimodal approach and state-of-the-art technology, this research project is designed to determine the prevalence, extent and nature of increased SNA in Asthma (AIM 1) and evaluate the impact of NHFT on sympathovagal balance in patients (AIM 2).

The project will address the following hypotheses:

1. SNA is increased in asthma patients.
2. NHFT has a positive impact on the sympathetic drive resulting in decreased SNA.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed Asthma
* Age ≥ 18
* Ability and willingness to give informed consent to participate in the study

Exclusion Criteria:

* Atrial fibrillation
* Active pacing of the heart by a cardiac pacemaker (i.e. no intrinsic heart rate)
* Clinically pre-established cardiovascular disease or other pulmonary diseases (e.g. arterial hypertension, systolic heart failure, COPD)
* In-patient stay in the hospital within the last 4 weeks prior to the study examination date
* Severe polyneuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthma patients (n=20) and Controls (n=10) patients without an established cardiovascular disease will be enrolled and the extent, nature and mechanism of SNA increase compared with healthy controls matched in a 2:1 ratio for age, sex and body mass index (BMI).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Assessments of the sympathetic nerve activity axis (Non invasive) | 1 year
  SVB (sympathovagal balance), HRV (Heart rate variability) and dBPV (diastolic blood pressure variability) will be analysed using a 3-lead electrocardiogram (sampling rate 1000Hz) and a continuous non-invasive arterial blood pressure signal (CNAP® technology, sampling rate 100Hz). HRV (ms2 based on continuously recorded variability in RR intervals) and (diastolic) BPV (expressed as mmHg2 based on continuously recorded variability in diastolic BP) will be computed by time domain analysis and by frequency domain analysis and presented as the high frequency component (HF; 0.15-0.4 Hz), low frequency component (LF; 0.04-0.15 Hz), their relative ratio low frequency/high frequency (LF/HF), and the very low frequency component (VLF; 0.0-0.04 Hz) for both HRV and dBPV .
  Outcome measure: LF/HF ratio of HRV.
Assessments of the sympathetic nerve activity axis (Invasive) | 1 year
  MSNA will be recorded via a tungsten microelectrode carefully placed in the peroneal nerve.
  Outcome measure: Burst Incidence (MSNA Bursts /100 beats).

SECONDARY OUTCOMES:
OSA severity | 1 year
  Outcome measure: Apnea-hypopnea Index/h (AHI /h; Scale 0 - 150 /h with higher values indicating more severe sleep apnea).
Determination of PH (pulmonary hypertension) and right HF (heart failure) severity | 1 year
  Outcome measure: TAPSE (tricuspid annular plane systolic excursion; mm).
Comprehensive lung function and inspiratory muscle function testing as previously described by our group | 1 year
  Outcome measure: Sniff nasal pressure (SNIP; cmH2O).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen-Department of Pneumology and Intensive Care, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spiesshoefer J, Becker S, Tuleta I, Mohr M, Diller GP, Emdin M, Florian AR, Yilmaz A, Boentert M, Giannoni A. Impact of Simulated Hyperventilation and Periodic Breathing on Sympatho-Vagal Balance and Hemodynamics in Patients with and without Heart Failure. Respiration. 2019;98(6):482-494. doi: 10.1159/000502155. Epub 2019 Aug 28. PMID 31461730
- [Background] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905
- [Background] Spiesshoefer J, Henke C, Herkenrath S, Brix T, Randerath W, Young P, Boentert M. Transdiapragmatic pressure and contractile properties of the diaphragm following magnetic stimulation. Respir Physiol Neurobiol. 2019 Aug;266:47-53. doi: 10.1016/j.resp.2019.04.011. Epub 2019 Apr 25. PMID 31029769
- [Background] Dysart K, Miller TL, Wolfson MR, Shaffer TH. Research in high flow therapy: mechanisms of action. Respir Med. 2009 Oct;103(10):1400-5. doi: 10.1016/j.rmed.2009.04.007. Epub 2009 May 21. PMID 19467849
- [Background] Bruni A, Garofalo E, Cammarota G, Murabito P, Astuto M, Navalesi P, Luzza F, Abenavoli L, Longhini F. High Flow Through Nasal Cannula in Stable and Exacerbated Chronic Obstructive Pulmonary Disease Patients. Rev Recent Clin Trials. 2019;14(4):247-260. doi: 10.2174/1574887114666190710180540. PMID 31291880
- [Background] Garrard CS, Seidler A, McKibben A, McAlpine LE, Gordon D. Spectral analysis of heart rate variability in bronchial asthma. Clin Auton Res. 1992 Apr;2(2):105-11. doi: 10.1007/BF01819665. PMID 1638105